CLINICAL TRIAL: NCT06309485
Title: An Open-Label Phase 2 Study of WGI-0301 Plus Sorafenib in Patients With Advanced Hepatocellular Carcinoma as Second Line Therapy
Brief Title: Phase 2 Study of WGI-0301 for Advanced HCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Haichang Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WGI0301-P2G-01
Record Dates: First submitted 2024-03-01; First posted 2024-03-13 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — Sorafenib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): WGI-0301 at MTD / RP2D dose with standard dose Sorafenib
  Interventions: Drug: WGI-0301 at MTD/RP2D dose IV infusion, QW; Drug: Sorafenib 400 mg PO, BID
- Arm B (Experimental): WGI-0301 at MTD / RP2D -1 dose with standard dose Sorafenib
  Interventions: Drug: WGI-0301 at MTD/RP2D -1 dose IV infusion, QW; Drug: Sorafenib 400 mg PO, BID continuously
- Arm C (Active Comparator): Standard dose Sorafenib alone
  Interventions: Drug: Sorafenib 400 mg PO, BID continuously

INTERVENTIONS:
Drug: WGI-0301 at MTD/RP2D dose IV infusion, QW — WGI-0301 is a lipid nanoparticle preparation of Archexin®, a 20-mer oligonucleotide that is complementary to Akt-1 mRNA, formulated for the treatment of advanced HCC.
  Arms: Arm A
Drug: WGI-0301 at MTD/RP2D -1 dose IV infusion, QW — WGI-0301 is a lipid nanoparticle preparation of Archexin®, a 20-mer oligonucleotide that is complementary to Akt-1 mRNA, formulated for the treatment of advanced HCC.
  Arms: Arm B
Drug: Sorafenib 400 mg PO, BID continuously — Sorafenib is an oral multi-kinase inhibitor used for the treatment of hepatocellular carcinoma.
  Arms: Arm B; Arm C
Drug: Sorafenib 400 mg PO, BID — Sorafenib is an oral multi-kinase inhibitor used for the treatment of hepatocellular carcinoma.
  Arms: Arm A

SUMMARY:
The purpose of this study is to determine the MTD of WGI-0301 in combination with Sorafenib for advanced Hepatocellular Carcinoma (HCC) and assess its safety and efficacy in adults with advanced unresectable HCC who have previously received PD-1 / PD-L1 immune checkpoint inhibitors.

DETAILED DESCRIPTION:
This study will include a two-stage design: Stage 1 (dose escalation) to determine the MTD/RP2D of WGI-0301 combined with Sorafenib. Stage 2 (dose expansion) with two different dose levels of WGI-0301 in combination with standard dose Sorafenib, or standard dose Sorafenib alone.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age on the day of signing informed consent, male or female.
2. Voluntarily agree to provide signed informed consent and are willing and able to comply with all aspects of the protocol.
3. Histologically or cytologically confirmed diagnosis of HCC. Diagnosis of HCC can be made without a biopsy if radiographic hallmarks of arterial hypervascularity and venous/ late phase washout are present by either dynamic contrast enhanced MRI or helical multidetector CT scan using contrast for a lesion > 2 cm, or by both modalities for a lesion 1~2 cm.
4. Barcelona Clinic Liver Cancer (BCLC) Stage C or BCLC stage B with bilobar involvement and infiltrative nature that is not amendable for local therapy (BCLC Classification see Appendix 7, Section 14.7).
5. Stage 1 only: At least first-line standard treatment failure (disease progression confirmed by imaging) or intolerance with no restriction on the number of prior lines of systemic treatment.
6. Stage 2 only: Patients must have objective radiographic disease progression or intolerance (Intolerance is defined as currently discontinued after ≥28 days of treatment due to toxicity) after only one prior line of systemic immunotherapy treatment with an anti-PD-1/ PD-L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies (Prior locoregional therapy such as surgery, radiofrequency ablation or trans-arterial chemoembolization are also allowed but not counted as systemic therapy, provided that progression has been documented after these therapies, and ≥4 weeks have elapsed since the last therapy).
7. Eligible for treatment with Sorafenib, as determined by investigators according to the Package Insert and clinical judgment.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1 within 7 days prior to the first dose of study intervention.
9. Patients must have at least one measurable lesion according to RECIST 1.1 as determined by the investigator, and that has not been the target of local or regional therapy including trans-arterial chemoembolization, intra-arterial chemotherapy, ethanol, or radiofrequency ablation; a new area of tumor progression within or adjacent to a previously treated lesion, if clearly measurable by a radiologist, is acceptable.
10. Stage 2 only: Patients must have at least one target lesion according to mRECIST that meet all the following criteria:

    * The lesion can be classified as a RECIST 1.1 measurable lesion.
    * The lesion is suitable for repeat measurement.
    * The lesion shows intratumoral arterial enhancement on contrast-enhanced CT or MRI.
11. Life expectancy in the judgement of the Investigator > 12 weeks.
12. Recovery to ≤ Grade 1 (CTCAE V5.0) from toxicities related to any prior treatments unless the adverse events are clinically non-significant and/ or stable with or without supportive therapy, except for alopecia (any grade) and Grade 2 peripheral neuropathy.
13. Collection of an archived tissue sample will be requested (where available) to support evaluation of the clinical utility of biomarker assessment in newly obtained vs. archived tissue samples; however, a subject will not be precluded from participating in the study if tissue sample is not available for collection or is otherwise insufficient for analysis.
14. Patients must have adequate organ function as defined below (Specimens must be collected within 7 days prior to the start of study intervention):

    * Child-Pugh Liver Function Class A (see Appendix 6 in Section 14.6)
    * AST or ALT ≤ 5.0 × ULN and total bilirubin ≤ 2 × ULN
    * Serum albumin ≥ 2.8 g/ dL
    * Creatinine Clearance (CrCL) ≥ 40 ml/ min (Cockcroft-Gault formula: CrCL (mL/ min) = [140-age(year)] × body weight (Kg)/ [72 × Scr (mg/ dl)]{ × 0.85 for female subjects})
    * International normalized ratio (INR) ≤ 2.0 (except for warfarin therapy)
    * Hemoglobin ≥ 8.5 g/ dL, absolute neutrophil count > 1000/ mm3, platelet count ≥ 60 000/ mm3 (no blood transfusion or blood products or granulocyte colony-stimulating factor within 14 days, corrected with erythropoietin or darbepoetin α are allowed)
15. Participants with hepatitis B virus (HBV) or hepatitis C virus (HCV) infection will be allowed if they meet the following criteria:

    * HBV-HCC: Resolved HBV infection (as evidenced by detectable HBV surface antibody, detectable HBV core antibody, undetectable HBV DNA, and undetectable HBV surface antigen) or chronic HBV infection (as evidenced by detectable HBV surface antigen or HBV DNA). Subjects with chronic HBV infection must have HBV DNA < 500 IU/ mL and must be on antiviral therapy. Active or uncontrolled clinically serious HBV infections are excluded.
    * HCV-HCC: Stable or resolved HCV infection (as evidenced by detectable HCV RNA or antibody).
16. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission per investigators' clinical judgment.
17. Women of child-bearing potential must have a negative urine or serum pregnancy within 3 days prior to receiving the first dose of study medication and must use accepted highly effective methods of contraception from the time of signing the informed consent through 6 months after the last dose of study drug. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, or be surgically sterile, for the duration of study participation, and for 3 months after completion of study drug administration. See Appendix 1 for protocol-approved highly effective methods of contraceptive combinations.

Exclusion Criteria:

1. Pregnant or breastfeeding patients or expecting to conceive or father children within the projected duration of the study.
2. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma.
3. Complete occlusion of the major portal vein or vena cava due to HCC (The major portal vein is defined as the part of portal vein between the union of the splenic and superior mesenteric veins and the first bifurcation into the left and right vein).
4. Major surgery within 4 weeks prior to the first dose of study intervention.
5. Previous identified allergy or hypersensitivity to components of WGI-0301 similar drugs or liposomal drugs or related excipients.
6. Previous identified allergy or hypersensitivity to components of Sorafenib or similar drugs.
7. Stage 2 only: Received prior Sorafenib therapy or any agents targeting AKT-PI3K pathway.
8. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of study intervention.
9. Locoregional therapy to liver within 6 weeks prior to the first dose, including but not limited to TACE, radiotherapy, radiofrequency ablation, microwave (except palliative radiotherapy for bone pain relief completed at least 2 weeks prior to the first dose).
10. Patients on concomitant use of strong CYP3A4 inducers (see Appendix 3 in Section 14.3) within 12 days prior to the first dose of study intervention. Additionally, patient in use of transporters based on FDA Drug Development and Drug Interactions, Table of Substrates, Inhibitors, and Inducers, or strong inducers of transporter, P-gp, including apalutamide, carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's wort. Patient in use of strong inhibitors of transporters based on based on FDA Drug Development and Drug Interactions, Table of Substrates, Inhibitors, and Inducers.
11. Clinically significant abnormalities of glucose metabolism (e.g., Patients with diabetes mellitus type1 or diabetes mellitus type 2 requiring treatment, or those with hemoglobin A1c (HbA1c) ≥8.0%.
12. clinically significant cardiovascular disease including:

    * Uncontrolled chronic hypertension defined as systolic > 150 mmHg or diastolic > 90 mmHg on more than one measurement despite optimal therapy (initiation or adjustment of BP medication prior to study entry is allowed provided that the average of 3 BP readings prior to enrollment is < 150/ 90 mmHg).
    * Hypotension as indicated by systolic blood pressure < 90 mmHg or mean arterial pressure < 65 mmHg on 2 consecutive measurements at the Screening Visit.
    * NYHA class III or IV Congestive heart failure, myocardial infarction or stroke, unstable angina pectoris, pericardial effusion (excluding trace pericardial effusion identified by echocardiography) or left ventricular ejection fraction < 45% within 6 months prior to the first dose.
    * Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, indeterminate cardiomyopathy).
    * Bradycardia (known history of cardiovascular disease and either physical examination at rest or electrocardiogram indicating heart rate < 50 bpm), or screening ECG indicating QTcF ≥ 470 msec, 2 retests at 30-minute intervals were required for the first abnormal QTcF, and 3 mean values were taken, Or there is severe arrhythmia requiring further treatment, including but not limited to ventricular fibrillation, atrial fibrillation, sustained ventricular tachycardia, second-degree or third-degree atrioventricular block, torsades de pointes, etc.
13. Clinically significant gastrointestinal disorders including:

    * Medical history of difficulty swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/ or absorption of the tested products
    * Gastrointestinal perforation and/ or fistula intra-abdominal abscess or intestinal obstruction within 6 months prior to the first dose
    * Clinically significant gastric bleeding within 6 months prior to the first dose (patients may be enrolled if esophageal and gastric varices are present on imaging, but no bleeding event or inpatient medical intervention occurs within 6 months prior to the first dose)
14. Clinically significant bleeding risks including:

    * Known hereditary or acquired bleeding or thrombotic tendencies (e.g., hereditary hemorrhagic telangiectasia or von Willebrand disease)
    * Bleeding symptoms such as hemoptysis (> 1/ 2 teaspoon bright red blood) and gastrointestinal bleeding within 3 months prior to screening
    * Thrombolytic agents within 10 days prior to the first dose
    * Receiving anticoagulant therapy (e.g., anticoagulants, antiplatelets) with an unstable anticoagulant regimen and/ or dosage (except sodium heparin for maintenance of central venous catheter patency)
15. History of solid organ transplant.
16. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
17. Known active or uncontrolled infection that could interfere with the study.
18. Uncontrolled ascites or pleural effusion requiring repeated drainage (investigator's judgment).
19. Past or current history of neoplasm other than HCC, except for curatively treated nonmelanoma skin cancer, in situ carcinoma of the cervix, or other cancer curatively treated and with no evidence of disease for at least 3 years.
20. Known central nervous system (CNS) or brain metastasis that is either symptomatic or untreated.
21. History of drug abuse or addiction at the present stage.
22. Subject has any other conditions or reason that, in the opinion of the Investigator, interferes with the ability of the subject to participate in the trial, places the subject at undue risk or complicates the interpretation of data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of WGI-0301 in combination with Sorafenib based on ORR per RECIST 1.1. | through study completion, an average of 2 year
  ORR is defined as the percentage of patients documented to have a confirmed CR or PR.

SECONDARY OUTCOMES:
Safety of each dose group. | through study completion, an average of 2 year
  Determined by number of AEs, SAEs, number of participant with changes in safety relevant clinical parameters, number of participants with dose modifications.
Tolerability of each dose group. | through study completion, an average of 2 year
  Determined by number of AEs, SAEs, number of participant with changes in safety relevant clinical parameters, number of participants with dose modifications.
Anti-tumor activity if WGI-0301 in combination with Sorafenib based on ORR. | through study completion, an average of 2 year
  ORR is defined as the percentage of patients documented to have a confirmed CR or PR.
Anti-tumor activity if WGI-0301 in combination with Sorafenib based on DCR. | through study completion, an average of 2 year
  DCR is defined as the percentage of patients documented to have a confirmed CR or PR or SD.
Anti-tumor activity if WGI-0301 in combination with Sorafenib based on DoR. | through study completion, an average of 2 year
  DoR is defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of objective PD or to death due to any cause in the absence of documented PD.
Anti-tumor activity if WGI-0301 in combination with Sorafenib based on PFS. | through study completion, an average of 2 year
  PFS is defined as the time from date of first study treatment to the date of PD or death (by any cause in the absence of progression) regardless of whether the patient withdraws from treatment or receives another anticancer therapy prior to progression.
Anti-tumor activity if WGI-0301 in combination with Sorafenib based on TTP per RECIST 1.1. | through study completion, an average of 2 year
  TTP is defined as the time from date of first study treatment to first documented PD.
Anti-tumor activity if WGI-0301 in combination with Sorafenib based on OS. | through study completion, an average of 2 year
  OS is defined as the time from date of first study treatment to death due to any cause.

IPD SHARING:
Plan to Share IPD: No